CLINICAL TRIAL: NCT03372356
Title: Psychosocial Screening for Neuroendocrine Tumor Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, MD, Professor, Chief of Department of GI Oncology, Peking University Cancer Hospital, Peking University
Other Study IDs: PSNET
Record Dates: First submitted 2017-12-10; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-08

CONDITIONS: Neuroendocrine Tumors
Keywords: DT; HADS; SPBS; CD-RISC; Psychosocial Screening
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neuroendocrine tumors: Patients with neuroendocrine tumors will be given access to an application that monitors distress, anxiety, depression, self-perceived burden, and resilience at regular intervals for 3 months lasting for 24 months.

SUMMARY:
This is a psychosocial screening application to usual care in a cohort of neuroendocrine tumor patients. The application involves monitoring using the NCCN Distress Thermometer(DT), Hospital Anxiety and Depression Scale(HADS), Self-Perceived Burden Scale(SPBS) and Connor-Davidson Resilience Scale(CD-RISC). These assessments will be completed at baseline, 3 months, 6 months, 12 months and 24 months. Patients will have the option of filling out questionnaires more frequently if desired.

ELIGIBILITY:
Inclusion Criteria:

1. sign written informed consent form;
2. age ≥ 18 years;
3. pathologically confirmed well-differentiated neuroendocrine tumors, G1-2 (Ki67≤20%);

Exclusion Criteria:

1. <18 years;
2. Neuroendocrine carcinoma;
3. History of psychiatric or psychologic illness;
4. History of previous cancers or cancer distress;
5. Patients with central nervous system(CNS) disorder；
6. Severe, uncontrolled medical condition that would affect patients' compliance;

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with well-differentiated neuroendocrine tumors, G1-2 (Ki67≤20%)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-08-09 (Actual); Primary Completion 2019-08-09 (Estimated); Study Completion 2020-08-09 (Estimated)

PRIMARY OUTCOMES:
DT | every 3 month until 24 month
  Distress Thermometer

SECONDARY OUTCOMES:
HADS | every 3 month until 24 month
  Hospital Anxiety and Depression Scale
SPBS | every 3 month until 24 month
  Self-Perceived Burden Scale
CD-RISC | every 3 month until 24 month
  Connor-Davidson Resilience Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No